CLINICAL TRIAL: NCT01013922
Title: A Descriptive Study to Explore Certain Characteristics of Patients at Risk for COPD in a Primary Care Setting
Brief Title: A Descriptive Study to Explore Certain Characteristics of Patients at Risk for Chronic Obstructive Pulmonary Disease (COPD) in a Primary Care Setting
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-RSE-DUM-2008/1
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; COPD-6; Spirometry; VC; FEV; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Patients with a smoking history of 15 pack years or more.

SUMMARY:
The purpose of this study is to explore if certain characteristics, easily detected within a regular primary care setting, may indicate that a patient at risk for COPD (45 ≤ age ≤ 80 years and a smoking history of ≥ 15 pack years) is prone to have a diagnosis of COPD according to Medical Products Agency guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of smoking one pack of cigarettes per day for 15 years or more

Exclusion Criteria:

* Known Chronic Obstructive Pulmonary Disease
* Known severe cardiovascular disease

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The patients will test their lung function with a COPD-6 screener for COPD and compare with regular spirometry. Medical records will be checked for health care contacts with respiratory diagnosis during the last 24 months prior to the study visit. | There will only be one visit in the study

CONTACTS AND LOCATIONS:
Overall Officials: Björn Tilling, Principal Investigator — Åtvidabergs vårdcentral; Georgios Stratelis, Study Director — AstraZeneca
Locations (23):
- Sweden (23):
  - Research Site, Alingsås
  - Research Site, Arvidsjaur
  - Research Site, Askim
  - Research Site, Åtvidaberg
  - Research Site, Bromma
  - Research Site, Eslöv
  - Research Site, Falun
  - Research Site, Gagnef
  - Research Site, Gothenburg
  - Research Site, Hagfors
  - Research Site, Helsingborg
  - Research Site, Hisings Kärra
  - Research Site, Höllviken
  - Research Site, Järpen
  - Research Site, Karlshamn
  - Research Site, Karlskrona
  - Research Site, Kil
  - Research Site, Limhamn
  - Research Site, Linköping
  - Research Site, Luleå
  - Research Site, Stockholm
  - Research Site, Timrå
  - Research Site, Värnamo

REFERENCES:
- [Derived] Thorn J, Tilling B, Lisspers K, Jorgensen L, Stenling A, Stratelis G. Improved prediction of COPD in at-risk patients using lung function pre-screening in primary care: a real-life study and cost-effectiveness analysis. Prim Care Respir J. 2012 Jun;21(2):159-66. doi: 10.4104/pcrj.2011.00104. PMID 22270480